CLINICAL TRIAL: NCT03116750
Title: Post-Market Clinical Follow-up Study with the ASPIREX®S Endovascular System to Assess the Safety and Effectiveness in the Treatment of DVT Patients and Special Patient Groups
Brief Title: Post-Market Clinical Follow-up Study with ASPIREX®S to Assess the Safety and Effectiveness in the Treatment of DVT
Acronym: P-MAX
Status: Completed | Type: Observational
Sponsor: Straub Medical AG (Industry)
Responsible Party: Sponsor
Other Study IDs: 15k013
Record Dates: First submitted 2017-03-31; First posted 2017-04-17 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Deep Vein Thrombosis; Bypass Complication; Dialysis Shunt; Stent Occlusion
Keywords: mechanical thrombectomy
MeSH Terms: conditions — Venous Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The ASPIREX®S Endovascular System is a rotating and aspirating catheter system. It is intended to be used for the percutaneous transluminal removal of fresh thrombotic or thromboembolic material from native blood vessels (or vessels fitted with stents, stent grafts or native or artificial bypasses) outside the cardiopulmonary, coronary and cerebral circulations.

CAPTUREX® , a catheter with a filter basket, is intended to be used for the filtering of emboli from blood vessels during potentially embolizing procedures on the patient.

ASPIREX®S and CAPTUREX® are CE-marked (Class III) medical devices. In this study the effectiveness and safety in the removal of thrombi in veins is assessed under real life setting.

ELIGIBILITY:
Inclusion Criteria:

1. Acute thrombotic or thromboembolic occlusion (onset of pain < 14 days)
2. Age > 18 years
3. Written informed consent form

Exclusion Criteria:

1. Patient not suitable for thrombectomy
2. Fracture area of broken stents
3. Known or suspected allergy to any of the components of the system or to a medicinal product to be administered in connection with the planned procedure
4. Persistent vasospasm
5. Severe coagulatory disorders
6. Patients with thrombophilia
7. Aneurysmatically altered vessel segments on target zone or on passage of catheter
8. Known or suspected infection, especially of the puncture site or the vessel segment being treated
9. Known, unhealed pre-existing mechanical damage to the vessel wall, especially caused by surgical procedures or interventional complications
10. Immature or not fully healed dialysis accesses or bypass grafts
11. Female subjects of childbearing capacity who are not willing to employ contraceptive measures
12. Pregnant or breast feeding subjects
13. Subjects who, in the opinion of the investigator, will be inappropriate for inclusion into this study or will not comply with requirements of the study
14. Subjects who are lawfully kept in an institution
15. Subjects who do not have the mental or physical ability to comply with time schedules and further study procedures
16. Current participation in any other clinical study (medicinal, medical device) or within the last 30 days prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Main study population: patients with DVT of the pelvis, legs and vena cava inferior.
  Additional patients with dialysis shunts and / or other bypasses, vena subclavia, vena brachiocephalica, vena cava superior, vena splenica and vena mesenterica superior/inferior will be included
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2024-06-06 (Actual)

PRIMARY OUTCOMES:
Procedural success (removal of occlusion and restoration of blood flow) | day of treatment
  Primary patency

SECONDARY OUTCOMES:
Adverse events | through study completion of 3 years
  failure of usability
Adverse device effects | through study completion of 3 years
  device related safety variables
Technical success rate | intraoperative
  removal of occlusion
Swelling of limb | through study completion of 3 years
  Circumference of the limb
Pain improvement | through study completion of 3 years
  pain disability index
additional Treatment , acute | before 72 hours after treatment
  index treatment at index site
additional Treatment, Long term | later than 72 hours after treatment
  index treatment at index site
Hospital Stay | 4-5 days after treatment
  Duration of hospital stay
Time to return back to ward | day of treatment
  Treatment time

CONTACTS AND LOCATIONS:
Locations (9):
- Austria (2):
  - Medizinische Universität Graz, Graz
  - Medizinische Universität Wien, Vienna
- CHU - Hôpital François-Mitterrand, Dijon, Bourgogne-Franche-Comté, France
- Germany (4):
  - Universitätsklinikum Aachen, Aachen
  - Klinikum Arnsberg, Klinik für Angiologie, Arnsberg
  - Universitätsklinikum Heidelberg, Heidelberg
  - Institut für Diagnostische und Interventionelle Radiologie, Universitätsklinik Rostock, Rostock
- Galway University Hospital, Galway, Ireland
- Azienda Ospedaliera San Giovanni Addolorata, Roma, Italy

IPD SHARING:
Plan to Share IPD: No